CLINICAL TRIAL: NCT00065169
Title: Anti-Inflammation in AD: PET Imaging Supplement
Brief Title: Delaying Alzheimer Disease Symptoms With Anti-Inflammatory Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Gary Small, MD, UCLA Professor of Psychiatry and Biobehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH058156 (NIH); R01MH058156 (NIH); DSIR AT-GP
Record Dates: First submitted 2003-07-17; First posted 2003-07-18 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Celecoxib

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
The purpose of this study is to determine whether the anti-inflammatory drug celecoxib can delay the onset of Alzheimer Disease (AD) in people with Age Associated Memory Impairment (AAMI). This study will also evaluate genetic risk and brain structure as potential predictors of mental decline.

DETAILED DESCRIPTION:
AD is one of the most common mental disorders of late life. Preliminary studies indicate that anti-inflammatory drugs may attenuate or prevent AD symptoms, but efficacy trials are needed.

Participants in this study will be randomly assigned to receive either celecoxib or placebo for 18 months. Participants will undergo positron emission tomography (PET) and magnetic resonance imaging (MRI) scans of the brain. Routine laboratory blood tests, cognitive tests, and an electrocardiogram (ECG) will be performed. Participants will also be screened for Parkinson disease. Follow-up testing will be conducted at specific intervals following the study.

ELIGIBILITY:
Inclusion Criteria:

* NIMH diagnostic criteria for Age Associated Memory Impairment (AAMI)
* Mini-Mental State Examination (MMSE) score between 26 and 30 (unless < 8 years of educational achievement)
* No significant cerebrovascular disease
* Estrogen replacement therapy and thyroid replacement therapy (if the participant is euthyroid) are permitted if the therapies are stable for > 1 month
* Memory and verbal fluency cut-off scores that increase the probability of incipient dementia (Buschke-Fuld: 34; verbal fluency: 46 for letters, 7 for categories; Benton Visual Retention: 5)
* Adequate visual and auditory acuity to allow neuropsychological testing
* Normal screening laboratory tests and electrocardiogram (ECG)

Exclusion Criteria:

* Possible or probable Alzheimer Disease (AD) or other dementia
* Neurologic or other physical illness that could produce cognitive deterioration
* History of transient ischemic attacks (TIAs), carotid bruits, or lacunes on an MRI scan
* History of myocardial infarction within the previous year or unstable cardiac disease
* Uncontrolled hypertension (systolic BP > 170 or diastolic BP > 100)
* History of significant liver disease, pulmonary disease, diabetes, or cancer
* DSM-IV criteria for major psychiatric disorders within the previous 2 years
* Past or present history of alcoholism or drug dependence
* Untreated depression as determined by a Hamilton Depression Rating Scale (HAM-D) score of 12 or more
* Drugs that may significantly affect psychometric test results
* Centrally active beta-blockers, narcotics, clonidine, anti-Parkinsonian medications, antipsychotics, benzodiazepines, systemic corticosteroids, medications with significant cholinergic or anticholinergic effects, anti-convulsants, warfarin, vitamins other than the standard multivitamin supplement, ginkgo biloba, and any nutraceuticals. Occasional chloral hydrate use will be allowed, but discouraged, for insomnia.
* Investigational drugs within the previous month or longer, depending on drug half-life
* Contraindication for MRI scan (e.g., metal in body, claustrophobia)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138
Dates: Start 2000-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Neuropsychiatric Institute, Los Angeles, California, United States